CLINICAL TRIAL: NCT00742053
Title: A Study of Electrocardiogram (ECG) Guidance for Placement of Peripherally Inserted Central Catheters (PICC)
Brief Title: Electrocardiogram (ECG) Guided Peripherally Inserted Central Catheter (PICC) Placement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment rate was too slow.
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Bard 3001
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-07

CONDITIONS: Primary Focus: Adult Subjects Who Require PICC Placement
Keywords: ECG PICC; Patients undergoing PICC placement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Male or female inpatients, age ≥ 18 and ≤ 80 years, who are in normal sinus rhythm and do not have a pacemaker or other indwelling intracardiac device and require PICC insertion for their routine care will be studied. Intervention: ECG-guided Power PICC placement.
  Interventions: Device: ECG-guided PICC placement

INTERVENTIONS:
Device: ECG-guided PICC placement — Patients undergoing PICC placement will have ECG data collected as a function of tip location.

SUMMARY:
This study is designed to obtain information for design purposes on use of an ECG guided monitoring system to aid in the correct placement of PICC lines.

There is no formal study hypothesis.

DETAILED DESCRIPTION:
PICC line placement is a common procedure, made more difficult by the need to ensure that catheter tip placement is in an acceptable location, typically the superior vena cava (SVC), and ideally at the junction of the SVC and right atrium. Tip location is determined at present by chest X-ray, which is performed after the procedure. If the tip location is incorrect, additional procedures and/or X-rays are needed until proper placement is ensured.

Use of an electrode placed inside the catheter during insertion has been reported to provide identifiable changes in the p-wave sufficient to guide placement. This study is designed to collect ECG and catheter depth information during routine PICC placement procedures, and to correlate these ECG changes to tip location as determined by contrast enhanced fluoroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Require Power PICC placement as standard care
* Signed informed consent

Exclusion Criteria:

* Has an intracardiac device
* Does not have normal sinus rhythm
* Has known abnormality of central venous system
* Plasma creatinine >=1.5 mg/dL
* Pregnancy
* Allergy or prior reaction to contrast material

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Michaels, MD, Principal Investigator — University of Utah Health Science Center
Locations (1):
- University of Utah Health Science Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith B, Neuharth RM, Hendrix MA, McDonnall D, Michaels AD. Intravenous electrocardiographic guidance for placement of peripherally inserted central catheters. J Electrocardiol. 2010 May-Jun;43(3):274-8. doi: 10.1016/j.jelectrocard.2010.02.003. Epub 2010 Mar 6. PMID 20206940

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at the University of Utah between August 2008 and December 2008.
Groups:
- PICC Insertion: All patients, aged 18 to 80 years, who required Peripherally inserted central catheter (PICC) insertion for their standard care will be studied.
Period: Overall Study
Arm/Group | PICC Insertion
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- PICC Insertion: All patients, aged 18 to 80 years, who required PICC insertion for their standard care will be studied.
Arm/Group | PICC Insertion
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.86 (15.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Distance of Maximum P-wave Amplitude in Relation to Superior Vena Cava (SVC)/Right Atrium(RA) Junction
Description: In order to determine correlation of PICC tip location with the intracatheter ECG, the PICC was advanced at 1cm increments and the p-wave observed for amplitude changes.
Time Frame: during catheter insertion
Measure: Mean (Standard Deviation); unit: cm
Groups:
- PICC Placement: Patients who require PICC placement
Arm/Group | PICC Placement
Number analyzed (Participants) | 6
cm | 0.5 (1.2)

ADVERSE EVENTS:
Time Frame: Subjects were followed for 1 day (about 24 hours) in order to verify and document the presence or absence of adverse events related to the study procedure
Arm/Group | PICC Insertion
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
The study was terminated early due to poor enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No